CLINICAL TRIAL: NCT05006417
Title: OnabotulinumtoxinA (Botox) Effect on Pain and Function in Recurrent Chronic Exertional Compartment Syndrome: a Pilot Study
Brief Title: Botox for the Treatment of Recurrent Chronic Exertional Compartment Syndrome
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: issues with supplier of strength testing equipment, presumed to go out of business
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-1375; Protocol Version 8/4/2021 (Other: UW Madison); A536120 (Other: UW Madison); SMPH/ORTHO&REHAB/REHAB MED (Other: UW Madison)
Record Dates: First submitted 2021-08-10; First posted 2021-08-16 (Actual); Results first posted 2024-07-18 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Compartment Syndrome of Leg
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Participants with R-CECS (Experimental): Botox to be injected under standard palpatory technique into the affected lower leg compartment.
  Interventions: Drug: Botox

INTERVENTIONS:
Drug: Botox — reconstituted at 100 units/mL, dosage will be based upon the affected muscles
  Other Names: OnabotulinumtoxinA

SUMMARY:
10 participants with Recurrent Chronic Exertional Compartment Syndrome (R-CECS) will be enrolled in a 6 month study at the University of Wisconsin Hospitals and Clinics to test the hypothesis that injection of Botox into the affected muscle group will alleviate pain associated with R-CECS.

DETAILED DESCRIPTION:
Participants will be enrolled in study at initial clinic visit by study staff at which time diagnosis of R-CECS will be established based on elevated pressure measurements in patients who have had surgical release of the affected compartments. Pressure testing will be performed outside of the clinical study and will be required to establish the diagnosis of R-CECS.

Initial clinic visit with study staff will consist of baseline measurements of ankle plantarflexion, dorsiflexion, inversion, and eversion strength using Kiio Force Sensor. The clinic visit with study staff will establish time point 0 and will consist of written consent for participation, Botox injection, and baseline University of Wisconsin Running Index (UWRI). Two months following this visit, the participant will have follow up with study staff. Study staff will again measure ankle strength (ankle inversion, eversion, plantarflexion, and dorsiflexion) using the Kiio Force Sensor utilizing the same strength assessment protocol. Study staff will monitor for side effects and administer the UWRI. Telephone follow up assessment of the UWRI will be made by study staff at 4 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Willing to provide written informed consent
* Willing to comply with all study procedures and be available for the duration of the study
* Documented diagnosis of R-CECS determined with elevated compartmental pressure testing following lower extremity fascia release (fasciotomy or fasciectomy)
* Females of childbearing potential must have a negative urine pregnancy test prior to enrollment and agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to randomization, for the duration of study participation, and for 7 days following completion of therapy.

  * A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

    * Has not undergone a hysterectomy or bilateral oophorectomy; or
  * Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).

Exclusion Criteria:

* History of hypersensitivity or allergy to any of the study drugs or drugs of similar chemical classes
* Known neuromuscular disease
* Known pulmonary disease including but not limited to asthma, pneumonia, or upper respiratory tract infection
* Dysphagia
* Known cardiac disease including but not limited to congestive heart failure, arrhythmia, or history of myocardial infarction
* Enrolled in another clinical trial or has used of any investigational drugs, biologics, or devices within 30 days prior to enrollment
* Currently or have taken in the past medications that affect neuromuscular function, aminoglycosides, muscle relaxants, or other botulinum neurotoxin agents. Currently taking any blood-thinning medications including, but not limited to Plavix, Coumadin, Eliquis, Xarelto
* Women who are pregnant or breast-feeding
* Vulnerable populations
* Not suitable for study participation due to other reasons at the discretion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-11-23 (Actual); Primary Completion 2022-11-23 (Actual); Study Completion 2022-11-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Suer, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One participant was enrolled in November of 2022
Period: Overall Study
Arm/Group | Participants With R-CECS
Started | 1
Baseline Measures | 1
2 Months | 0
4 Months | 0
6 Months | 0
Completed | 0
Not Completed | 1
Not completed — PI terminated study for problems with strength testing equipment | 1

BASELINE CHARACTERISTICS:
Arm/Group | Participants With R-CECS
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Score
Description: Change in pain score (0-10, where 10 is increased pain) will be assessed at each time point will be assessed at each time point (2, 4, 6 months) using Friedman's ANOVA.
Time Frame: 2 months, 4 months, 6 months
Population: only baseline data collected before study was terminated
Groups:
- Participants With R-CECS - Left Leg; Participants With R-CECS - Right Leg: Botox to be injected under standard palpatory technique into the affected lower leg compartment.
  Botox: reconstituted at 100 units/mL, dosage will be based upon the affected muscles
Arm/Group | Participants With R-CECS - Left Leg | Participants With R-CECS - Right Leg
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Number of Participants With Lower Extremity Weakness
Description: A primary safety endpoint is incidence of lower extremity weakness, measured by
Time Frame: up to 6 months
Population: study terminated early
Arm/Group | Participants With R-CECS
Number analyzed (Participants) | 0

3. Primary Outcome: Incidence of Adverse Events
Description: A primary safety endpoint is the incidence of adverse events, such as bruising, bleeding, pain, redness, or swelling where the injection was given.
Time Frame: one study visit (within 2 hours)
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With R-CECS
Number analyzed (Participants) | 1
Participants | 0

4. Secondary Outcome: Change in Ankle Dorsiflexion Strength Using Kiio Force Sensor
Description: A Kiio Force Sensor will be used to measure the change in ankle strength. Change in strength outcomes at baseline and 2 months will be assessed using Wilcoxon signed rank tests or, if necessary, linear mixed effects models for repeated measures, to account for intra-subject correlation (left and right legs).
Time Frame: baseline and month 2
Population: strength equipment not functional, study terminated as a result
Measure: Number; unit: pounds of force
Arm/Group | Participants With R-CECS - Left Leg | Participants With R-CECS - Right Leg
Number analyzed (Participants) | 1 | 1
pounds of force
  baseline | 24.9 | 25.2
  2 months: number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change in Ankle Plantarflexion Strength Using Kiio Force Sensor
Description: as for outcome 4
Time Frame: baseline and month 2
Population: strength equipment not functional, study terminated as a result
Measure: Number; unit: pounds of force
Arm/Group | Participants With R-CECS - Left Leg | Participants With R-CECS - Right Leg
Number analyzed (Participants) | 1 | 1
pounds of force
  baseline | 154.3 | 156.4
  2 months: number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change in Ankle Inversion Strength Using Kiio Force Sensor
Description: as for outcome 4
Time Frame: baseline and month 2
Population: strength equipment not functional, study terminated as a result
Measure: Number; unit: pounds of force
Arm/Group | Participants With R-CECS - Left Leg | Participants With R-CECS - Right Leg
Number analyzed (Participants) | 1 | 1
pounds of force
  baseline | 22.9 | 22.8
  2 months: number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change in Ankle Eversion Strength Using Kiio Force Sensor
Description: as for outcome 4
Time Frame: baseline and month 2
Population: strength equipment not functional, study terminated as a result
Measure: Number; unit: pounds of force
Arm/Group | Participants With R-CECS - Left Leg | Participants With R-CECS - Right Leg
Number analyzed (Participants) | 1 | 1
pounds of force
  baseline | 22.7 | 22.8
  2 months: number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Change in Ability to Perform Activities of Daily Living
Description: A question on the University of Wisconsin Running Index (UWRI) asks the participant to indicate how their running injury impacts their ability to perform daily activities. The scoring is on a 5 point likert scale from 0 = unable to perform, 1 = significantly impact, 2 = moderately impact, 3 = slightly impact, to 4 = no impact.
Time Frame: baseline, 2 months, 4 months, 6 months
Population: study was terminated after baseline measure
Measure: Number; unit: score on a scale
Arm/Group | Participants With R-CECS
Number analyzed (Participants) | 1
score on a scale
  baseline | 2
  2 months: number analyzed (Participants) | 0
  4 months: number analyzed (Participants) | 0
  6 months: number analyzed (Participants) | 0

9. Secondary Outcome: Participant Frustration With Injury
Description: A question on the UWRI asks the participant to indicate how frustrated they are by their running injury. The scoring is on a 5 point likert scale from 0 = extremely frustrated, 1 = significantly frustrated, 2 = moderately frustrated, 3 = mildly frustrated, to 4 = not frustrated.
Time Frame: baseline, 2 months, 4 months, 6 months
Population: study was terminated after baseline measure
Measure: Number; unit: score on a scale
Arm/Group | Participants With R-CECS
Number analyzed (Participants) | 1
score on a scale
  baseline | 0
  2 months: number analyzed (Participants) | 0
  4 months: number analyzed (Participants) | 0
  6 months: number analyzed (Participants) | 0

10. Secondary Outcome: Participant Perception of Recovery From Injury
Description: A question on the UWRI asks the participant to indicate how much recovery have they made from their running injury. The scoring is on a 5 point likert scale from 0 = no recovery, 1 = minimal recovery, 2 = moderate recovery, 3 = significant recovery, to 4 = complete recovery.
Time Frame: baseline, 2 months, 4 months, 6 months
Population: study was terminated after baseline measure
Measure: Number; unit: score on a scale
Arm/Group | Participants With R-CECS
Number analyzed (Participants) | 1
score on a scale
  baseline | 0
  2 months: number analyzed (Participants) | 0
  4 months: number analyzed (Participants) | 0
  6 months: number analyzed (Participants) | 0

11. Secondary Outcome: Pain in the 24 Hours Following Running
Description: A question on the UWRI asks the participant to indicate how much pain they experience during the 24 hours following a run. The scoring is on a 5 point likert scale from 0 = unable to run, 1 = significant pain, 2 = moderate pain, 3 = minimal pain, to 4 = no pain.
Time Frame: baseline, 2 months, 4 months, 6 months
Population: study was terminated after baseline measure
Measure: Number; unit: score on a scale
Arm/Group | Participants With R-CECS
Number analyzed (Participants) | 1
score on a scale
  baseline | 0
  2 months: number analyzed (Participants) | 0
  4 months: number analyzed (Participants) | 0
  6 months: number analyzed (Participants) | 0

12. Secondary Outcome: Change in Running Duration: Weekly
Description: A question on the UWRI asks the participant to indicate if their weekly mileage or weekly running time changed as a result of their injury. The scoring is on a 5 point likert scale from 0 = unable to run, 1 = significantly reduced, 2 = moderately reduced, 3 = minimally reduced, to 4 = same or greater than before my injury.
Time Frame: baseline, 2 months, 4 months, 6 months
Population: study was terminated after baseline measure
Measure: Number; unit: score on a scale
Arm/Group | Participants With R-CECS
Number analyzed (Participants) | 1
score on a scale
  baseline | 0
  2 months: number analyzed (Participants) | 0
  4 months: number analyzed (Participants) | 0
  6 months: number analyzed (Participants) | 0

13. Secondary Outcome: Change in Running Duration: Longest Run
Description: A question on the UWRI asks the participant to indicate if the distance of their longest weekly run has changed as a result of their injury. The scoring is on a 5 point likert scale from 0 = unable to run, 1 = significantly reduced, 2 = moderately reduced, 3 = minimally reduced, to 4 = same or longer than before my injury.
Time Frame: baseline, 2 months, 4 months, 6 months
Population: study was terminated after baseline measure
Measure: Number; unit: score on a scale
Arm/Group | Participants With R-CECS
Number analyzed (Participants) | 1
score on a scale
  baseline | 0
  2 months: number analyzed (Participants) | 0
  4 months: number analyzed (Participants) | 0
  6 months: number analyzed (Participants) | 0

14. Secondary Outcome: Change in Running Speed
Description: as for outcome 13
Time Frame: baseline, 2 months, 4 months, 6 months
Population: study was terminated after baseline measure
Measure: Number; unit: score on a scale
Arm/Group | Participants With R-CECS
Number analyzed (Participants) | 1
score on a scale
  baseline | 0
  2 months: number analyzed (Participants) | 0
  4 months: number analyzed (Participants) | 0
  6 months: number analyzed (Participants) | 0

15. Secondary Outcome: Participant Confidence in Increasing the Duration and Intensity of Running
Description: A question on the UWRI asks the participant to indicate how their injury affects their confidence to increase the duration or intensity of their running. The scoring is on a 5 point likert scale from 0 = I cannot increase my running, 1 = if I increase, I might get worse, 2 = neutral, 3 = if I increase I might be fine, to 4 = confident to increase my running.
Time Frame: baseline, 2 months, 4 months, 6 months
Population: study was terminated after baseline measure
Measure: Number; unit: score on a scale
Arm/Group | Participants With R-CECS
Number analyzed (Participants) | 1
score on a scale
  baseline | 0
  2 months: number analyzed (Participants) | 0
  4 months: number analyzed (Participants) | 0
  6 months: number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: one study visit (within 2 hours)
Arm/Group | Participants With R-CECS
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-09): https://cdn.clinicaltrials.gov/large-docs/17/NCT05006417/Prot_SAP_000.pdf